CLINICAL TRIAL: NCT01178944
Title: Pralatrexate in Combination With Oxaliplatin in Advanced Esophago-gastric Cancer: A Phase II Trial With Predictive Molecular Correlates
Brief Title: Pralatrexate and Oxaliplatin in Treating Patients With Unresectable or Metastatic Esophageal, Stomach, or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 169210; NCI-2010-01583 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 169210 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2010-08-09; First posted 2010-08-10 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Esophageal Undifferentiated Carcinoma; Gastric Adenocarcinoma; Gastric Squamous Cell Carcinoma; Recurrent Esophageal Adenocarcinoma; Recurrent Esophageal Squamous Cell Carcinoma; Recurrent Gastric Carcinoma; Stage IIIB Esophageal Adenocarcinoma; Stage IIIB Esophageal Squamous Cell Carcinoma; Stage IIIB Gastric Cancer; Stage IIIC Esophageal Adenocarcinoma; Stage IIIC Esophageal Squamous Cell Carcinoma; Stage IIIC Gastric Cancer; Stage IV Esophageal Adenocarcinoma; Stage IV Esophageal Squamous Cell Carcinoma; Stage IV Gastric Cancer; Undifferentiated Gastric Carcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma; Stomach Neoplasms | interventions — Oxaliplatin; 10-propargyl-10-deazaaminopterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pralatrexate, oxaliplatin) (Experimental): Patients receive pralatrexate IV over 3-5 minutes and oxaliplatin IV over 2 hours on day 1. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity. Oxaliplatin will be discontinued after 12 courses.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Oxaliplatin; Drug: Pralatrexate

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Drug: Pralatrexate — Given IV
  Other Names: 10-propargyl-10-deazaaminopterin; Folotyn; PDX

SUMMARY:
This phase II trial studies how well pralatrexate and oxaliplatin work in treating patients with esophageal, stomach, or gastroesophageal junction cancer that cannot be removed by surgery or has spread from the primary site (place where it started) to other places in the body. Pralatrexate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pralatrexate with oxaliplatin may be an effective treatment for esophageal, stomach, or gastroesophageal junction cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall response rate in patients with advanced esophago-gastric cancer (EGC) to combination pralatrexate and oxaliplatin.

SECONDARY OBJECTIVES:

I. To examine the toxicity and tolerability of this regimen. II. To determine the time-to-progression and overall survival using this regimen.

III. To examine whether functionally relevant polymorphisms of genes of the folate metabolism pathway correlate with efficacy and toxicity of pralatrexate.

IV. To examine whether response to pralatrexate can be predicted by micro-ribonucleic acid (microRNA) expression profiling of the epithelial component of the tumor.

OUTLINE:

Patients receive pralatrexate intravenously (IV) over 3-5 minutes and oxaliplatin IV over 2 hours on day 1. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity. Oxaliplatin will be discontinued after 12 courses.

After completion of study treatment, patients are followed up for 30 days and then periodically thereafter for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed carcinoma of the esophagus, stomach or gastro-esophageal junction that is metastatic, or locally advanced and inoperable for cure; histological sub-types permitted include adenocarcinoma, squamous-cell carcinoma, or undifferentiated carcinoma; small-cell carcinoma variant is not eligible
* No previous systemic therapy for metastatic or recurrent disease; therapy (chemotherapy, radiotherapy, or both) administered in the neo-adjuvant, adjuvant, or definitive setting for previously localized disease is permitted, provided it was completed more than 6 months prior to enrollment; palliative radiotherapy is permitted provided it is completed >= 3 weeks prior to study therapy initiation
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy >= 12 weeks
* Hemoglobin >= 9 g/dl
* Absolute neutrophil count >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Serum creatinine =< institutional upper limit normal (ULN)
* Bilirubin =< 1.5 x ULN
* Transaminases =< 3 x ULN; for documented liver metastases, transaminases up to 5 x ULN is permitted
* No evidence of >= grade 2 peripheral neuropathy
* Patients with reproductive potential must be willing to use an adequate contraceptive method (e.g., abstinence, intrauterine device, oral contraceptives, barrier device with spermicide or surgical sterilization) during treatment and for three months after completing treatment; a negative pregnancy test is required for women of child-bearing potential; nursing women are ineligible
* Written, informed consent

Exclusion Criteria:

* Hypersensitivity to platinum compounds
* Uncontrolled inter-current illness including but not limited to active infection, symptomatic congestive heart failure, unstable angina, uncontrolled cardiac arrhythmia, or psychiatric illness that would limit compliance with study requirements
* Presence of brain metastases
* Patients with third-space (pleural, peritoneal) fluid not controllable with usual drainage methods are not eligible
* History of second primary malignancy within 3 years prior to enrollment, except for in-situ cervix carcinoma or non-melanoma skin cancer
* Undergone an allogeneic stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-09; Primary Completion 2015-01 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Khushalani, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Rochester General Hospital, Rochester, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Pralatrexate, Oxaliplatin)
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Treatment (Pralatrexate, Oxaliplatin)
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate to combination pralatrexate and oxaliplatin as assessed by Response Evaluation Criteria in Solid Tumors version 1.1. Objective responses will be confirmed 4 weeks after first documentation of response. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 5 years
Population: All Cohort -1 treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Pralatrexate, Oxaliplatin)
Number analyzed (Participants) | 31
percentage of participants | 26 [12 to 45]

2. Secondary Outcome: Number of Participants With an Adverse Event
Description: Number of participants with an adverse event. Please refer to the adverse event reporting for more detail. Incidence of toxicity as assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0
Time Frame: Up to 30 days after the last dose of study drug(s)
Population: All treated and eligible patients
Measure: Number; unit: participants
Arm/Group | Treatment (Pralatrexate, Oxaliplatin)
Number analyzed (Participants) | 35
participants | 35

3. Secondary Outcome: Overall Survival (OS)
Description: Estimated using the Kaplan-Meier method and proportional hazards models.
Time Frame: From the date of study enrollment to the time of death from any cause, assessed up to 5 years
Population: All treated and eligible patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pralatrexate, Oxaliplatin)
Number analyzed (Participants) | 35
months | 7.2 [6.4 to 10.8]

4. Secondary Outcome: Time to Progression (TTP)
Description: Estimated using the Kaplan-Meier method and proportional hazards models.
Time Frame: From the date of study enrollment to the first observation of progressive disease, assessed up to 5 years
Population: All treated and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pralatrexate, Oxaliplatin)
Number analyzed (Participants) | 35
months | 5.1 [3.4 to 6.4]

5. Other Pre Specified Outcome: Overall Survival (OS) for SNP ATIC/AICART - s10932606 Genotypes
Description: Kaplan-Meier estimates of median survival time for each genotype
Time Frame: From the date of study enrollment up to 5 years
Population: All treated and eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pralatrexate, Oxaliplatin)
Number analyzed (Participants) | 35
months
  C: number analyzed (Participants) | 24
  C | 10.22 [6.74 to 12.39]
  T: number analyzed (Participants) | 4
  T | 18.71 [2.33 to 31.38]
  TC: number analyzed (Participants) | 7
  TC | 4.63 [2.30 to 5.45]

6. Other Pre Specified Outcome: MicroRNA Expression - miR-215-5p
Description: Mean microRNAs expression of mi-215-5p in tumor tissues of responders and non-responders using a microfabricated device called a gene chip.
Time Frame: Baseline
Population: All treated participants that had enough tissue to perform microdissection to collect epithelial cells for subsequent microRNA profiling.
Measure: Mean (95% Confidence Interval); unit: Arbitrary fluorescent intensity
Arm/Group | Treatment (Pralatrexate, Oxaliplatin)
Number analyzed (Participants) | 29
Arbitrary fluorescent intensity
  Responders: CR+PR | 6.6 [5.7 to 7.1]
  Non responders: stable disease/progression | 5.6 [5.3 to 5.9]
Statistical Analysis 1: Comparison: Treatment (Pralatrexate, Oxaliplatin); Comparison is CR+PR vs stable disease/progression; Test type: Other; p = 0.585, t-test, 2 sided; Mean Difference (Final Values) = 1.08, 95% CI 2-sided [0.78 to 1.38]

ADVERSE EVENTS:
Arm/Group | Treatment (Pralatrexate, Oxaliplatin)
Serious Adverse Events (participants affected / at risk) | 10/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pralatrexate, Oxaliplatin) (N=35)
Myocardial infarction (Cardiac disorders) | 1 (2)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 1 (2)
Disease progression (General disorders) | 1 (2)
Pyrexia (General disorders) | 1 (2)
Infection (Infections and infestations) | 1 (4)
Lung infection (Infections and infestations) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (2)
Haemoglobin (Investigations) | 1 (4)
Dehydration (Metabolism and nutrition disorders) | 3 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Haemorrhage intracranial (Nervous system disorders) | 1 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pralatrexate, Oxaliplatin) (N=35)
Anaemia (Blood and lymphatic system disorders) | 9 (37)
Leukopenia (Blood and lymphatic system disorders) | 12 (65)
Lymphopenia (Blood and lymphatic system disorders) | 12 (32)
Neutropenia (Blood and lymphatic system disorders) | 12 (42)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (50)
Tachycardia (Cardiac disorders) | 3 (6)
Dry eye (Eye disorders) | 1 (4)
Eye discharge (Eye disorders) | 2 (4)
Eye pain (Eye disorders) | 1 (2)
Lacrimation increased (Eye disorders) | 1 (2)
Vision blurred (Eye disorders) | 2 (6)
Abdominal pain (Gastrointestinal disorders) | 7 (16)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (6)
Ascites (Gastrointestinal disorders) | 1 (4)
Constipation (Gastrointestinal disorders) | 13 (42)
Diarrhoea (Gastrointestinal disorders) | 14 (71)
Dry mouth (Gastrointestinal disorders) | 3 (6)
Dyspepsia (Gastrointestinal disorders) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 6 (20)
Faecal incontinence (Gastrointestinal disorders) | 1 (2)
Flatulence (Gastrointestinal disorders) | 1 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (2)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (2)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 22 (96)
Odynophagia (Gastrointestinal disorders) | 1 (2)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (2)
Oesophagitis (Gastrointestinal disorders) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 30 (169)
Vomiting (Gastrointestinal disorders) | 17 (55)
Asthenia (General disorders) | 1 (2)
Chest pain (General disorders) | 4 (8)
Chills (General disorders) | 1 (2)
Early satiety (General disorders) | 1 (2)
Fatigue (General disorders) | 23 (103)
Gait disturbance (General disorders) | 1 (2)
Infusion site extravasation (General disorders) | 1 (2)
Localised oedema (General disorders) | 1 (2)
Oedema (General disorders) | 1 (2)
Oedema peripheral (General disorders) | 8 (25)
Pain (General disorders) | 1 (2)
Pyrexia (General disorders) | 3 (6)
Temperature intolerance (General disorders) | 3 (10)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (8)
Hypersensitivity (Immune system disorders) | 3 (6)
Abdominal wall infection (Infections and infestations) | 1 (2)
Infection (Infections and infestations) | 1 (4)
Nasopharyngitis (Infections and infestations) | 1 (2)
Oral candidiasis (Infections and infestations) | 2 (4)
Oral infection (Infections and infestations) | 1 (2)
Pneumonia (Infections and infestations) | 1 (2)
Skin infection (Infections and infestations) | 1 (4)
Upper respiratory tract infection (Infections and infestations) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (2)
Feeding tube complication (Injury, poisoning and procedural complications) | 1 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (2)
Thermal burn (Injury, poisoning and procedural complications) | 1 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (2)
Alanine aminotransferase increased (Investigations) | 2 (10)
Aspartate aminotransferase (Investigations) | 5 (16)
Aspartate aminotransferase increased (Investigations) | 12 (40)
Blood alkaline phosphatase (Investigations) | 6 (15)
Blood alkaline phosphatase increased (Investigations) | 9 (27)
Blood creatinine (Investigations) | 4 (10)
Blood creatinine increased (Investigations) | 2 (3)
Carbon dioxide increased (Investigations) | 1 (2)
Haemoglobin (Investigations) | 12 (75)
Haemoglobin decreased (Investigations) | 9 (47)
Lymphocyte count decreased (Investigations) | 9 (49)
Neutrophil count decreased (Investigations) | 5 (13)
Platelet count decreased (Investigations) | 5 (21)
Weight decreased (Investigations) | 14 (42)
White blood cell count decreased (Investigations) | 6 (18)
Decreased appetite (Metabolism and nutrition disorders) | 9 (25)
Dehydration (Metabolism and nutrition disorders) | 8 (16)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 7 (21)
Hypernatraemia (Metabolism and nutrition disorders) | 4 (8)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 18 (69)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (6)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (8)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (27)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (10)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (9)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (8)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (2)
Dizziness (Nervous system disorders) | 6 (16)
Dizziness postural (Nervous system disorders) | 1 (2)
Dysaesthesia (Nervous system disorders) | 2 (4)
Dysgeusia (Nervous system disorders) | 11 (24)
Headache (Nervous system disorders) | 6 (11)
Neuropathy peripheral (Nervous system disorders) | 1 (2)
Paraesthesia (Nervous system disorders) | 4 (22)
Peripheral sensory neuropathy (Nervous system disorders) | 27 (106)
Peroneal nerve palsy (Nervous system disorders) | 1 (4)
Sinus headache (Nervous system disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 2 (6)
Confusional state (Psychiatric disorders) | 1 (2)
Delirium (Psychiatric disorders) | 1 (2)
Hallucination (Psychiatric disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (4)
Restlessness (Psychiatric disorders) | 1 (2)
Chromaturia (Renal and urinary disorders) | 1 (2)
Dysuria (Renal and urinary disorders) | 1 (2)
Haematuria (Renal and urinary disorders) | 1 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (2)
Pollakiuria (Renal and urinary disorders) | 2 (3)
Urinary incontinence (Renal and urinary disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (10)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (8)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 (24)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (4)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 6 (12)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (2)
Medical diet (Surgical and medical procedures) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 5 (10)
Embolism (Vascular disorders) | 1 (2)
Hot flush (Vascular disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (2)
Hypotension (Vascular disorders) | 5 (10)
Orthostatic hypotension (Vascular disorders) | 1 (2)
Superior vena cava syndrome (Vascular disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT01178944/Prot_SAP_000.pdf